CLINICAL TRIAL: NCT05459818
Title: Individual Patient Data Meta-Analysis of Prospective Studies of Patients Treated With the GORE® VIABAHN® Endoprosthesis With Heparin Bioactive Surface (VSX) for Peripheral Arterial Disease (INSIGHT VSX)
Brief Title: Individual Patient Data Analysis of Viabahn for Peripheral Arterial Disease
Acronym: Insight-VSX
Status: Completed | Type: Observational
Sponsor: Rijnstate Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-2052
Record Dates: First submitted 2022-07-06; First posted 2022-07-15 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Peripheral Vascular Diseases
Keywords: peripheral artarial disease; endovascular treatment; endoprosthesis; Viabahn; Individual patient data analysis
MeSH Terms: conditions — Peripheral Vascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Viabahn implanted — An individual patient data analysis obtained from databases used in prospective studies that published results of patients treated with the latest generation heparin-bonded Viabahn in the femoropopliteal artery.
  Other Names: endovascular treatment

SUMMARY:
To evaluate the effectiveness of the VSX device in pre-determined patient populations to understand the patient characteristics that impact outcomes.

DETAILED DESCRIPTION:
Rationale: Studies on the efficacy of self-expanding covered stents for the treatment of patients with superficial femoral artery (SFA) occlusive disease have mainly focused on stent patency. Subgroup analysis was often not feasible, related to small sample sizes. This pooled analysis of individual patient-level data provides larger sample sizes and a more heterogeneous population, which allows for the ability to perform subgroup analyses to identify patients that will most benefit from VSX treatment. The current analysis will provide insights into the effectiveness of the VSX device for specific subgroups.

Objective: To evaluate the effectiveness of the VSX device in pre-determined patient populations to understand the patient characteristics that impact outcomes.

Study design: Multicenter retrospective individual patient data meta-analysis. Study population: Patients treated with a VSX device for de novo or restenotic lesions of the superficial femoral artery and previously enrolled in a prospective VSX study whom were treated for SFA disease with the latest generation heparin-bonded Viabahn, and published in peer reviewed journals.

Main study parameters/endpoints: The primary study parameter is primary patency at 12-months. In addition, for all subjects and for subgroups as described further below, the following secondary endpoints will be evaluated through follow-up: primary patency at 24 months, primary assisted patency, secondary patency, freedom from Target Lesion Revascularization (TLR) at 12 and 24 months, clinical Improvement, minor and major amputation, mortality. The following subgroup analysis will be performed if sufficient data are available: critical limb threatening ischemia patients (Rutherford 4-6), patients with intermittent claudication (Rutherford 1-3), chronic total occlusions, by gender, by number of runoff vessels, lesion length, TASC II lesion classification, calcified lesions, by device diameter.

ELIGIBILITY:
Inclusion Criteria:

1. Patient was enrolled and treated with the GORE® VIABAHN® Endoprosthesis with Heparin Bioactive Surface device in a Gore-sponsored or physician-sponsored study for de novo or restenotic lesions of the femoropopliteal artery.
2. Lesions ≥10 cm in length and TASC C or D classification will be included
3. Patient-level data can be obtained and pooled with other studies

Exclusion Criteria:

1. Patient was not formally enrolled in their corresponding study (e.g., training cases)
2. Patient was enrolled for treatment of in-stent restenotic lesions.
3. Patient has incomplete or missing data that does not allow for analysis.
4. Case reports (n<10 patients)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: An individual patient data analysis obtained from databases used in prospective studies that published results of patients treated with the latest generation heparin-bonded Viabahn in the femoropopliteal artery. For this purpose authors are asked to provide extensive patient information (anonymized): patient characteristics at baseline (e.g. comorbidities), lesion details, procedural details, hospitalization details, follow-up visits.
Sampling Method: Non-Probability Sample
Enrollment: 977 (Actual)
Dates: Start 2022-10-12 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
Primary patency | at 12 months.
  Primary patency is defined as no evidence of restenosis or occlusion within the originally treated lesion based on color-coded duplex sonography (CDUS, PSVR < 2.5) or no angiographic evidence of stenosis > 50% if CDUS is uninterpretable or unavailable.

SECONDARY OUTCOMES:
Primary patency | at 24 months
  Primary patency is defined as no evidence of restenosis or occlusion within the originally treated lesion based on color-coded duplex sonography (CDUS, PSVR < 2.5) or no angiographic evidence of stenosis > 50% if CDUS is uninterpretable or unavailable.
Primary assisted patency | 12 and 24 months
  Primary assisted patency is defined as flow through the treated lesion with or without repeat percutaneous intervention completed prior to complete vessel occlusion.
Secondary patency | 12 and 24 months
  Secondary patency is defined as patency in the target lesion maintained by repeat intervention after complete occlusion of the treated arterial segment.
Freedom from Target Lesion Revascularization (TLR) | 12 and 24 months
  Freedom from revascularization of the treated lesion after either restenosis or occlusion by means of a percutaneous vascular intervention, surgical by-pass, thrombolysis, or other such invasive means.
Clinical Improvement | 12 and 24 months
  Clinical improvement is defined as at least one-group improvement in Rutherford Classification compared to baseline.
Major amputation | 12 and 24 months
  Surgical removal of a portion of the study limb (generally above the ankle, transmetatarsal, or metatarsal)
Mortality | 12 and 24 months
  Death, overall and procedure-related (until 30 days)

CONTACTS AND LOCATIONS:
Overall Officials: MMPJ Reijnen, Prof, Principal Investigator — Rijnstate
Locations (1):
- Rijnstate, Arnhem, Netherlands

IPD SHARING:
Plan to Share IPD: No
On request data can be shared with other researchers after publication of the data; consent needs to be collected from all collaborators